CLINICAL TRIAL: NCT03250507
Title: Mixture of Liposomal Bupivicaine and Bupivicaine Hydrogen Chloride (HCl) May Provide Faster and Longer Lasting Analgesia in Transversus Abdominis Block for Patient Having Open Abdominal Hysterectomies
Brief Title: Mixture of Liposomal Bupivacaine and Bupivacaine for TAP Block for Open Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Mohamed Rida Alsaden, Anesthesiologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 10655
Record Dates: First submitted 2017-04-05; First posted 2017-08-15 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Hysterectomy
Keywords: TAP block; Liposomal bupivicaine
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of three study groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, surgical team, nursing team, anesthesia team, and outcomes assessor will be blinded to the group assignment. The anesthetist performing the TAP block will not be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bupivacaine (Active Comparator): Patients will receive a TAP block with 60 mL 0.25% bupivacaine. this group will not receive Liposomal bupivacaine
  Interventions: Drug: Bupivacaine
- Liposomal bupivacaine (Active Comparator): Patients will receive a TAP block with 20 mL liposomal bupivacaine and 40 mL saline.
  this group will not receive bupivacaine. they receive only liposomal bupivacaine.
  Interventions: Drug: Liposomal bupivacaine; Drug: Saline
- Liposomal bupivacaine and bupivacaine (Experimental): Patients will receive a TAP block with 20 mL liposomal bupivacaine and 40 mL 0.25% bupivacaine.
  this group will receive the mixture of Liposomal bupivacaine and bupivacaine.
  Interventions: Drug: Bupivacaine; Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 0.25% bupivacaine for TAP block
  Other Names: Marcaine, Sensorcaine
  Arms: Bupivacaine; Liposomal bupivacaine and bupivacaine
Drug: Liposomal bupivacaine — Exparel for TAP block
  Other Names: Exparel
  Arms: Liposomal bupivacaine; Liposomal bupivacaine and bupivacaine
Drug: Saline — Saline for TAP block that will be mixed with liposomal bupivacaine to bring the liposomal bupivacaine group to 60 mL total volume.
  Arms: Liposomal bupivacaine

SUMMARY:
The goal of this study is to evaluate the effectiveness of different formulations of bupivacaine infiltrated into the transversus abdominis plane (TAP) on post-operative pain management after open abdominal hysterectomy.

DETAILED DESCRIPTION:
All eligible patients who consent to the study will be randomized to one of three groups. Group 1 will receive a TAP block with 60 mL 0.25% bupivacaine. Group 2 will receive a TAP block with 20 mL liposomal bupivacaine and 40 mL saline. Group 3 will receive a TAP block with 20 mL liposomal bupivacaine and 40 mL 0.25% bupivacaine. Patients will be assessed in the post-anesthesia care unit (PACU) at once each on Post-operative day 1,2, and 3.

ELIGIBILITY:
Inclusion Criteria:

* Elective open abdominal hysterectomy with midline incision, age > 18 years, American Society of Anesthesiologist classification score (ASA classification) 1-3.

Exclusion Criteria:

* Patient with a chronic pain condition, major unexpected surgical complication, unexpected prolonged intubation, patient refusal, local anesthetic allergy, any contraindication to regional anesthesia, greater than 2 attempts by resident and greater than 1 attempt by staff anesthesiologist for TAP block.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible patients are undergoing open abdominal hysterectomy and therefore are female.
Enrollment: 90 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed-Rida Alsaden, MBChB FRCPC, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will be available to only study researchers.

REFERENCES:
- [Derived] Fidkowski CW, Choksi N, Alsaden MR. A randomized-controlled trial comparing liposomal bupivacaine, plain bupivacaine, and the mixture of liposomal bupivacaine and plain bupivacaine in transversus abdominus plane block for postoperative analgesia for open abdominal hysterectomies. Can J Anaesth. 2021 Jun;68(6):773-781. doi: 10.1007/s12630-020-01911-1. Epub 2021 Jan 11. PMID 33432496

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine: Patients will receive a TAP block with 20 mL liposomal bupivacaine and 40 mL saline.
  this group will not receive bupivacaine. they receive only liposomal bupivacaine.
  Liposomal bupivacaine: Exparel for TAP block
  Saline: Saline for TAP block that will be mixed with liposomal bupivacaine to bring the liposomal bupivacaine group to 60 mL total volume.
- Liposomal Bupivacaine and Bupivacaine: Patients will receive a TAP block with 20 mL liposomal bupivacaine and 40 mL 0.25% bupivacaine.
  this group will receive the mixture of Liposomal bupivacaine and bupivacaine.
  Bupivacaine: 0.25% bupivacaine for TAP block
  Liposomal bupivacaine: Exparel for TAP block
Period: Overall Study
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 13 patients were excluded from study analysis due to meeting exclusion criteria. N=25 in group Bupi, N = 27 in group Liposomal bupi, and N=25 in group liposomal bupi and bupi. 20 patients were discharged within 72 hr. Data is given for those in the hospital for 24 hr periods. For the period 24-48 hr, n = 24 in group bupivacaine, n = 26 in group liposomal, n = 25 in group mixture. For the period 48-72 hr, n = 18 for group bupivacaine, n = 20 for group liposomal, and n = 19 for group mixture. *
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 90
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 30 | 90
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption During the First 72 Hours Postoperatively as Measured in Morphine Equivalents (mg)
Description: Total opioid consumption
Time Frame: 0 - 72 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 18 | 20 | 19
mg morphine equivalents | 208 [155 to 270] | 203 [153 to 283] | 202 [116 to 325]

2. Primary Outcome: Time to First Opioid Consumption as Measured in Hours Until the First Dose of Breakthrough Opioid Medication Given
Description: time to first opioid given
Time Frame: 0 - 72 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 25 | 27 | 25
minutes | 51 [28 to 66] | 63 [44 to 102] | 51 [24 to 84]

3. Secondary Outcome: Patient Satisfaction Using 3 Point Scale - Very Satisfied, Satisfied, Not Satisfied
Description: Patient satisfaction post-operatively. The number of patients who were very satisfied is reported.
Time Frame: 0 - 72 hours post-operatively
Measure: Number; unit: participants
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 25 | 27 | 25
participants | 9 | 13 | 9

4. Secondary Outcome: Length of Stay in the Hospital
Description: Length of stay in the hospital, maximum time until discharge from the hospital
Time Frame: until the patient is discharged from the hospital
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 25 | 27 | 25
hours | 79 [61 to 122] | 82 [72 to 102] | 80 [76 to 107]

5. Secondary Outcome: Number of Patients With Local Anesthetic Toxicity
Description: Presence of local anesthetic toxicity
Time Frame: 0 - 72 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 25 | 27 | 25
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With Hypotension < 60 mmHg Mean Arterial Pressure
Description: Presence of hemodynamic instability
Time Frame: 0 - 72 hours post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 25 | 27 | 25
Participants | 0 | 1 | 5

7. Secondary Outcome: Pain Scores Using Visual Analogue Scale ( 0-10)
Description: Maximum pain score 0 - 24 hr. Pain scores are reported on a scale of 0-10. 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, and 7-10 = severe pain.
Time Frame: 0-24 postoperative pain scores
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
Number analyzed (Participants) | 25 | 27 | 25
units on a scale | 8 [7 to 9] | 7 [6 to 7] | 7 [5 to 8]

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Liposomal Bupivacaine and Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03250507/Prot_SAP_001.pdf